CLINICAL TRIAL: NCT05785481
Title: Early Neurological Outcome in Newborns With Mild Encephalopathy:a Regional Network
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Romeo Domenico Marco, Assistant professor, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2631
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Hypoxic Encephalopathy
Keywords: Mild Hypoxic Encephalopathy
MeSH Terms: conditions — Hypoxia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with early diagnosis (within 6 hours of life) of mild HIE
  Interventions: Diagnostic Test: Clinical and instrumental neurological assessment

INTERVENTIONS:
Diagnostic Test: Clinical and instrumental neurological assessment — During the neonatal period:
  neurological objective exam according to the modified Sarnat score, Thompson score and Hammersmith Neonatal Neurological Examination (HINE) within 6 hours of life, 24 hours of life and before resignation; an AEEG study within 6 hours of life, for 6 hours; cerebral ultrasound within 6 hours of life, in the third and seventh day of life; a brain magnetic resonance imaging study between the seventh and 14th day of life; an EEG evaluation within 7 days.
  After resignation, all patients will be included in a minimum duration follow-up program of 12 months, with assessments at 3rd, 6th and 12th month of age:
  Hammersmith Neonatal Neurological Examination (HINE) and evaluation of the General Movements; evaluation of psychomotor development through Griffiths/Bayley III scales at the 12th month; EEG evaluation at the 6th and 12th month.

SUMMARY:
This is a multicenter prospective observational study that aims to determine the natural history of patients with early diagnosis (within 6 hours of life) of mild hipoxic ischemic encephalopaty (HIE), who are not candidates for treatment with therapeutic hypothermia. The goal of this study is to learn about the early neurological outcome in babies with mild encephalopathy, as recent studies have shown how there is an increased risk of brain damage with a high incidence of resonance magnetic nuclear (RMN) anomalies and possible neurodevelopmental complications including learning or neuropsychological disorders, epilepsy, visual and sensory deficits. The main question aimed to answer is the identification of early possible predictive factors for an unfavorable outcome in order to undertake early rehabilitation programs and for the future planning of trials on early neuroprotection in the investigated population. Babies with early diagnosis (within 6h of life) of mild grade HIE not candidate for hypothermic treatment are subjected to clinical and instrumental assessments during the neonatal period:

* neurological objective exam according to the modified "Sarnat" score, Thompson score and Hammersmith Neonatal Neurological Examination (HINE) within 6 hours of life, 24 hours of life and before resignation;
* an Amplitude Electroencephalogram (aEEG) study within 6 hours of life, for 6 hours;
* cerebral ultrasound within 6 hours of life, in the third and seventh day of life;
* a brain magnetic resonance imaging study between the seventh and 14th day of life;
* an Electroencephalogram (EEG) evaluation within 7 days.

After resignation, all patients will be included in a minimum duration follow-up program of 12 months, with assessments at 3rd, 6th and 12th month of age:

* Hammersmith Neonatal Neurological Examination (HINE) and evaluation of the General Movements;
* evaluation of psychomotor development through Griffiths/Bayley III scales at the 12th month;
* EEG evaluation at the 6th and 12th month.

ELIGIBILITY:
Inclusion Criteria:

* patients born after the 36th week of gestational age, with signs of encephalopathy found between the 10th minute of life and 6h, presenting with one or more of the following signs of intrapartum hypoxia with a potential of hydrogeb (pH) ≤ 7 or an excess of bases (BE) ≥ 12 mmol/l in the first hour of life, measured on cord or arterial blood or an abnormal course of delivery (eg: fetal heart rate abnormalities, cord prolapse, uterine tear, haemorrhage/ trauma/ convulsive seizures/ maternal cardiorespiratory arrest; shoulder dystocia; meconium-dyed amniotic fluid or protracted second stage and the presence of an Apgar at 10 min ≤5 or the need for continuous respiratory support at 10 minutes.

Exclusion Criteria:

* mutes neurological objectivity;
* impossibility of recruitment within 6h;
* major congenital anomalies, brain malformations;
* neonatal abstinence syndrome;
* metabolic encephalopathies and severe growth restriction (birth weight ≤1800g);
* treatment with therapeutic hypothermia;
* refusal of consent.

Ages: 10 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with early diagnosis (within 6 hours of life) of mild HIE, who are not candidates for treatment with therapeutic hypothermia
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
early neurological outcome | between the seventh and 14th day of life
  the percentage of patients with mild asphyxia with evidence of brain damage, defined by MRI
early neurological outcome | at the 6th month
  the percentage of patients with mild asphyxia with evidence of brain damage, defined by EEG abnormalities
early neurological outcome | at 12th month.
  the percentage of patients with mild asphyxia with evidence of brain damage, defined by EEG abnormalities
early neurological outcome | at the 3th month
  the percentage of patients with mild asphyxia with evidence of brain damage, defined by neurological examination
early neurological outcome | at the 6th month.
  the percentage of patients with mild asphyxia with evidence of brain damage, defined by neurological examination
early neurological outcome | at the 12th month.
  the percentage of patients with mild asphyxia with evidence of brain damage, defined by neurological examination

SECONDARY OUTCOMES:
Electroencephalographic and epilepsy outcome | between the 6 hours of life and 12th month.
  percentage of abnormalities at electroencephalographic checks and presence of critical events
Neurodevelopmental outcome | 12th month
  percentage of abnormalities at Neurodevelopmental evaluation
Hospitalization | between birth until 12th month
  Duration of Hospitalization
adverse events | between birth until 12th month
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Domenico M Romeo, MD,PHD, Principal Investigator — ChatolicUIT
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli -IRRCS, Rome, Italy